CLINICAL TRIAL: NCT03115359
Title: A Comparative Effectiveness Randomized Controlled Trial of Mindfulness Meditation Versus Cognitive Behavioral Therapy for Opioid-Treated Chronic Low Back Pain
Brief Title: Strategies to Assist With Management of Pain
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0353; A532007 (Other: UW, Madison); SMPH/FAMILY MED/FAMILY MED (Other: UW, Madison); Protocol_V20-00, 03.07.2022 (Other: HS-IRB UW, Madison)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Opioid Therapy; Chronic Pain; Mindfulness Meditation; Cognitive Behavioral Therapy; Opioid-treated Chronic Low Back Pain; CLBP
MeSH Terms: conditions — Chronic Pain | interventions — Meditation; Mindfulness; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness randomized controlled trial of two behavioral interventions
Who Masked: Investigator
Masking Description: Although participants, therapists and outcome assessors cannot be blinded to the study intervention, investigators and analysts will be blinded to the group status until the first stages of analysis and reporting are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Therapy (Experimental): Mindfulness Based Therapy intervention, adjunctive to usual care for opioid-treated chronic low back pain.
  Interventions: Behavioral: Mindfulness Based Therapy
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy intervention, adjunctive to usual care for opioid-treated chronic low back pain.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Therapy — The Mindfulness Based Therapy intervention will teach participants the mindfulness meditation-based strategies, tailored to the needs of those with opioid-treated chronic lower back pain. It consists of eight weekly 2-hour group sessions guided by trained therapists. In addition to session attendance, participants are asked to practice at home at least 6 days/week, 30 minutes/day during the study.
  In addition to the intervention, the participants will receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
  Other Names: Meditation; Mindfulness Meditation; Mindfulness
  Arms: Mindfulness Based Therapy
Behavioral: Cognitive Behavioral Therapy — The Cognitive Behavioral Therapy (CBT) intervention will teach participants the CBT-based strategies, tailored to the needs of those with opioid-treated chronic lower back pain. It consists of eight weekly 2-hour group sessions guided by trained therapists. In addition to session attendance, participants are asked to practice at home at least 6 days/week, 30 minutes/day during the study.
  In addition to the intervention, the participants will receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Chronic low back pain (CLBP) has no known effective treatment. While often treated with long-term opioid therapy, opioids do not work well for many patients and can cause serious side effects, including addiction, poorer mental health, and overdose death. Even when paired with a standard-of-care cognitive behavioral therapy (CBT), results are limited. Patients, families and clinicians are very interested in using alternative treatments for CLBP, especially complementary and integrative treatments such as mindfulness meditation (MM). MM helps train the mind to bring non-judgmental and accepting attention to present-moment experiences such as pain. MM offers an active and safe self-care approach to chronic pain that contrasts with the passive and potentially harmful nature of opioid treatment, and may prove more effective than CBT in helping improve health and well-being, and reduce reliance on opioids in adults with opioid-treated CLBP. Although this hypothesis is supported by early research, including a pilot study by the Principal Investigator, evidence on MM's effectiveness in this population is inconclusive, presenting a critical knowledge gap.

With input from patients, family members, and clinicians, the Investigators have designed a study to address this gap and propose a clinical trial that will compare the effectiveness of MM to standard-of-care CBT in opioid-treated CLBP. Based on the existing research, it is hypothesized that MM training will lead to a larger reduction in pain intensity, increase in physical function, improvement in quality of life, and decrease in daily opioid dose, as compared to CBT training, with benefits of MM especially notable in adults with worse mood, anxiety or unhealthy opioid-use behaviors who often experience more severe symptoms of CLBP and less improvement in response to existing therapies.

To test these hypotheses, 766 adults with opioid-treated CLBP will be randomly assigned into one of two 8-week treatment groups: MM (383 participants) that will receive the MM training or CBT (383 participants) that will receive the CBT training. Due to the COVID-19 pandemic-related restrictions, the study protocol was modified in October 2020 so that the study can be completed virtually.

The effectiveness of MM versus CBT will be assessed over a 12-month period with patient-reported measures, recommended by experts and endorsed by our stakeholder partners, including patients with opioid-treated CLBP, their families and clinicians.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is the most common disabling chronic noncancer pain condition treated with opioids. Many opioid-treated patients experience inadequate pain relief and disability as well as dose-dependent adverse effects of opioids, such as worse mental health, opioid misuse, overdose and death. They frequently have co-occurring depression, anxiety, and opioid use disorders, which worsen outcomes. Poor outcomes and opioid-related harms underscore the need for safe and effective strategies for chronic pain care and opioid dose reduction, especially in high-impact, opioid-treated pain, as noted by the Institute of Medicine, the National Institutes of Health, and the Patient-Centered Outcomes Research Institute.

The investigators pilot randomized controlled trial (RCT) of mindfulness meditation (MM), a popular mind-body modality, demonstrated its potential to safely improve the health of patients and reduce opioid dosage in opioid-treated CLBP. To expand the evidence for MM for use in opioid-treated chronic pain, the investigators propose a 5-year multi-site, mixed-methods pragmatic RCT comparing the effectiveness of MM to standard-of-care cognitive behavioral therapy (CBT) for improving outcomes in opioid-treated CLBP. The study team will follow 766 participants over 12 months and compare outcomes that matter to patients and their families in 383 adults randomized to the MM group to 383 adults randomized to the CBT group, controlling for relevant factors.

The specific aims of this study are:

1. To compare the effectiveness of MM to CBT for reducing pain and increasing function. Current study is based on hypothesis that adults with opioid-treated CLBP in the MM group will report a greater reduction in pain severity and a greater increase in function at 6 and 12 months compared to those in the CBT group.
2. To compare the effectiveness of MM to CBT for improving quality of life (QoL) and reducing daily opioid dose. Study team hypothesize that adults with opioid-treated CLBP in the MM group will report a greater improvement in QoL and a greater decrease in daily opioid dose at 6 and 12 months compared to those in the CBT group.
3. To examine if participant baseline characteristics impact treatment response to MM or CBT. Study team hypothesize that among those with increased baseline symptom severity of negative affect (anxiety, depression) and opioid misuse behaviors, MM will be more beneficial than CBT for improving Aim 1 and Aim 2 outcomes.

Both MM and CBT interventions are patterned after established programs, adapted to meet the needs of patients with opioid-treated CLBP, with input from content experts and patient partners. The manualized interventions are delivered by trained therapists over 8 weeks in weekly two-hour group sessions in addition to care the participants are already receiving from their regular clinicians; during the COVID-19 pandemic, the interventions are delivered virtually. Participants are also be asked to practice MM or CBT strategies at home during the entire study (at least 30 minutes/day, 6 days/week).

Eligibility criteria will focus on English-speaking adults ≥21 years old, with moderate-to-severe CLBP treated with ≥15 mg/day of morphine-equivalent opioid dose for ≥3 months. The study will implement a limited set of exclusionary criteria to ensure a diverse sample, from which findings can be generalized.

Outcome measures were selected and prioritized based on guidelines and stakeholder input. They are collected at baseline, at 3, 6, 9 and 12 months. Only baseline and 12 months post-entry data collection is conducted in person; the 3, 6, and 9-month data collection occurs online or by phone to minimize burden. Due the COVID-19 pandemic, the study protocol was modified to allow for the completion of all assessments and data collection virtually.

Pain severity and function, as assessed by standard, validated survey measures, will serve as primary (Aim 1), and quality of life and opioid dose (morphine-equivalent mg/day) as secondary (Aim 2) outcomes. Severity of negative affect (depression, anxiety) and opioid misuse behaviors, also measured by validated surveys, are the main hypothesized predictors of treatment success (Aim 3). The repeated measures intention-to-treat outcome analysis will compare the change in primary and secondary outcomes over the 12 month period and across the two groups. To determine prognostic factors of treatment effect, a linear mixed model analysis will be performed for Aim 1 and Aim 2 outcomes, adjusting for potential confounders, study site and a random intercept for subject.

A team of experienced investigators and engaged stakeholders will carry out this multi-health system, multi-site study led by the faculty from the University of Wisconsin (Madison, WI), Harvard Medical School (Boston, MA) and the University of Utah (Salt Lake City, UT). Stakeholders helped develop this proposal and will be integrally involved as partners in all aspects of the study, from finalizing the methods, trouble-shooting implementation of the research plan, and dissemination of results.

Positive findings of this study could help improve health outcomes and reduce daily opioid dose in patients with opioid-treated CLBP, and inform clinical decisions of patients and clinicians about the choice between MM and CBT for opioid-treated CLBP.

*The Results Reporting due date has been extended per PCORI to be 9/30/2023.

ELIGIBILITY:
Inclusion Criteria (per self-report): English-speaking; age ≥ 21 years old; chronic low back pain (defined as a pain in lumbosacral region or sciatica for ≥3 months), with an average daily back pain score ≥3 on a 0-10 numerical rating scale (question from the Brief Pain Inventory), treated with ≥30 mg/day of morphine-equivalent dose for ≥3 months; at least moderate CLBP-related disability (≥21 score on the Oswestry Disability Index); capable of giving informed consent; willing to complete the study activities.

Exclusion Criteria (per self-report): prior formal Mindfulness Meditation or Cognitive Behavioral Therapy training; current pregnancy; diagnosis of borderline personality, delusional, or bipolar (mania) disorder; inability to safely or reliably participate in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra E Zgierska, MD PhD, Principal Investigator — Penn State University; Bruce P Barrett, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries, programming codes, qualitative codebooks, and other study materials will be provided to the funding agency, Patient-Centered Research Outcomes Institute (PCORI) after the study completion in order to promote replication of the research process. A final, clean dataset will be available for data sharing after the project and analysis completion. PCORI may share these materials and data upon request, after consultation with the PI.

REFERENCES:
- [Derived] Zgierska AE, Edwards RR, Barrett B, Burzinski CA, Jamison RN, Nakamura Y, Henningfield MF, Tuan WJ, Shen C, Sehgal N, Lennon RP, Dong H, Chinchilli VM, Liu Y, Turnquist A, Schiefelbein AR, Jacobs EA, Veasley C, Cowan P, Garland EL. Mindfulness vs Cognitive Behavioral Therapy for Chronic Low Back Pain Treated With Opioids: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e253204. doi: 10.1001/jamanetworkopen.2025.3204. PMID 40193079
- [Derived] Zgierska AE, Burzinski CA, Garland EL, Lennon RP, Jamison R, Nakamura Y, Barrett B, Sehgal N, Mirgain SA, Singles JM, Cowan P, Woods D, Edwards RR. Mindfulness-based therapy compared to cognitive behavioral therapy for opioid-treated chronic low back pain: Protocol for a pragmatic randomized controlled trial. Contemp Clin Trials. 2021 Nov;110:106548. doi: 10.1016/j.cct.2021.106548. Epub 2021 Sep 1. PMID 34478870
- See also: Strategies To Assist with Management of Pain (STAMP) Study Website — http://www.STAMPstudy.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Based Therapy: Mindfulness Based Therapy intervention, adjunctive to usual care for opioid-treated chronic low back pain.
  Mindfulness Based Therapy: The Mindfulness Based Therapy intervention will teach participants the mindfulness meditation-based strategies, tailored to the needs of those with opioid-treated chronic lower back pain. It consists of eight weekly 2-hour group sessions guided by trained therapists. In addition to session attendance, participants are asked to practice at home at least 6 days/week, 30 minutes/day during the study.
  In addition to the intervention, the participants will receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy intervention, adjunctive to usual care for opioid-treated chronic low back pain.
  Cognitive Behavioral Therapy: The Cognitive Behavioral Therapy (CBT) intervention will teach participants the CBT-based strategies, tailored to the needs of those with opioid-treated chronic lower back pain. It consists of eight weekly 2-hour group sessions guided by trained therapists. In addition to session attendance, participants are asked to practice at home at least 6 days/week, 30 minutes/day during the study.
  In addition to the intervention, the participants will receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
Period: Overall Study
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Started | 385 | 385
Completed | 266 | 263
Not Completed | 119 | 122
Not completed — Withdrawal by Subject | 29 | 39
Not completed — Scheduling conflict | 25 | 23
Not completed — Personal reasons including health | 12 | 9
Not completed — Transportation barriers | 3 | 0
Not completed — No longer interested | 5 | 4
Not completed — No reason provided | 45 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 385 | 385 | 770
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.9) | 58.0 (11.7) | 57.8 (11.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 233 | 201 | 434
  Male | 147 | 181 | 328
  missing, declined, unknown, unspecified | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Not Hispanic or Latino | 316 | 331 | 647
  Unknown or Not Reported | 52 | 36 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 33 | 37 | 70
  White | 307 | 310 | 617
  More than one race | 13 | 9 | 22
  Unknown or Not Reported | 26 | 20 | 46
Composite Pain Severity [Mean (Standard Deviation); unit: score on a scale] — Averaged 4 pain severity items from the Brief Pain Inventory (0-10 scale; higher indicates higher level of pain)
  score on a scale | 6.0 (1.4) | 6.2 (1.5) | 6.1 (1.5)
Physical Function [Mean (Standard Deviation); unit: score on a scale] — 10-item Oswestry Disability Index (0-100 scale; higher score indicates higher level of back pain-related functional limitation)
  score on a scale | 47.3 (13.6) | 47.0 (14.3) | 47.2 (14.0)
Health-Related Quality of Life (Physical Health) [Mean (Standard Deviation); unit: score on a scale] — 12-item Short Form-12 (0-100 scale; higher score indicates better physical health function)
  score on a scale | 28.8 (8.1) | 28.2 (8.5) | 28.5 (8.3)
Health-Related Quality of Life (Mental Health) [Mean (Standard Deviation); unit: score on a scale] — 12-item Short Form-12 (0-100 scale; higher score indicates better mental health function)
  score on a scale | 41.6 (11.1) | 43.3 (12.4) | 42.5 (11.8)
Average Daily Opioid Dose [Mean (Standard Deviation); unit: morphine-MG equivalent dose per day] — Timeline Followback Method (morphine-MG equivalent dose [mg/day] over the prior 14 days). Log transformation was required because of the skewed distribution of the daily opioid dose data in the primary effectiveness analysis.
  morphine-MG equivalent dose per day | 163 (601) | 191 (1344) | 177 (1041)
Negative Affect [Mean (Standard Deviation); unit: score on a scale] — 14-item Hospital Anxiety and Depression Scale (0-42 scale; higher score indicates more negative affect)
  score on a scale | 16.7 (7.2) | 16.2 (8.0) | 16.4 (7.6)
Negative Affect [Count of Participants; unit: Participants] — 14-item Hospital Anxiety and Depression Scale (0-42 scale; higher score indicates more negative affect). HADS scores >11 points have been associated with worse treatment outcomes in individuals with opioid-treated chronic pain.
  Participants
    Score greater than 11 | 289 | 261 | 550
    Score less than or equal to 11 | 96 | 123 | 219
    Missing | 0 | 1 | 1
Opioid Use Behaviors [Mean (Standard Deviation); unit: score on a scale] — 17-item Current Opioid Misuse Measure (0-68 scale; higher score indicates more opioid use behaviors)
  score on a scale | 9.2 (6.4) | 10.0 (7.4) | 9.6 (6.0)
Opioid Use Behaviors [Count of Participants; unit: Participants] — 17-item Current Opioid Misuse Measure (0-68 scale; higher score indicates more opioid use behaviors). COMM scores ≥9 points have been linked to increased risk for opioid misuse, OUD, anxiety and depression.
  Participants
    scores greater than or equal to 9 | 174 | 175 | 349
    scores less than 9 | 209 | 207 | 416
    Missing | 2 | 3 | 5
Average Pain Severity [Mean (Standard Deviation); unit: score on a scale] — 1 'average' pain severity item from the Brief Pain Inventory (0-10 scale; higher score indicates higher level of pain)
  score on a scale | 6.0 (1.5) | 6.2 (1.7) | 6.1 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Composite Pain Severity
Description: Averaged 4 pain severity items from the Brief Pain Inventory (0-10 scale; higher indicates higher level of pain)
Time Frame: 6 months post-entry
Population: Number of participants analyzed varies due to some participants not providing data for a given measure(s). Reasons for missing data include participants declining to answer a particular question/survey, participant withdrawals, lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 253 | 227
score on a scale | 5.6 (1.7) | 5.6 (1.8)

2. Primary Outcome: Composite Pain Severity
Description: Averaged 4 pain severity items from the Brief Pain Inventory (0-10 scale; higher indicates higher level of pain)
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 249 | 232
score on a scale | 5.5 (1.8) | 5.5 (1.9)

3. Primary Outcome: Physical Function
Description: 10-item Oswestry Disability Index (0-100 scale; higher score indicates higher level of back pain-related functional limitation)
Time Frame: 6 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 250 | 226
score on a scale | 44.6 (16.1) | 45.1 (16.4)

4. Primary Outcome: Physical Function
Description: as for outcome 3
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 249 | 232
score on a scale | 43.4 (15.3) | 43.2 (15.4)

5. Primary Outcome: Average Pain Severity
Description: 1 'average' pain severity item from the Brief Pain Inventory (0-10 scale; higher score indicates higher level of pain)
Time Frame: 6 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 253 | 227
score on a scale | 5.6 (1.7) | 5.5 (1.9)

6. Primary Outcome: Average Pain Severity
Description: 1 'average' pain severity item from the Brief Pain Inventory (0-10 scale; higher score indicates higher level of pain)
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 249 | 232
score on a scale | 5.4 (1.9) | 5.5 (2.0)

7. Secondary Outcome: Health-Related Quality of Life (Physical Health)
Description: 12-item Short Form-12 (0-100 scale; higher score indicates better physical health function)
Time Frame: 6 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 250 | 226
score on a scale | 30.7 (8.7) | 29.9 (9.4)

8. Secondary Outcome: Health-Related Quality of Life (Physical Health)
Description: 12-item Short Form-12 (0-100 scale; higher indicates better physical health function)
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 248 | 232
score on a scale | 30.5 (8.8) | 30.0 (9.2)

9. Secondary Outcome: Health-Related Quality of Life (Mental Health)
Description: 12-item Short Form-12 (0-100 scale; higher score indicates better mental health function)
Time Frame: 6 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 250 | 226
score on a scale | 43.2 (11.4) | 43.5 (12.1)

10. Secondary Outcome: Health-Related Quality of Life (Mental Health)
Description: 12-item Short Form-12 (0-100 scale; higher score indicates better mental health function)
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 248 | 232
score on a scale | 43.5 (11.5) | 45.9 (11.0)

11. Secondary Outcome: Average Daily Opioid Dose
Description: Timeline Followback Method (morphine-MG equivalent dose [mg/day] over the prior 14 days). Log transformation was required because of the skewed distribution of the daily opioid dose data in the primary effectiveness analysis.
Time Frame: 6 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: morphine-MG equivalent dose per day
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 269 | 250
morphine-MG equivalent dose per day | 119 (521) | 191 (1603)

12. Secondary Outcome: Average Daily Opioid Dose
Description: as for outcome 11
Time Frame: 12 months post-entry
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: morphine-MG equivalent dose per day
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 253 | 237
morphine-MG equivalent dose per day | 144 (556) | 192 (1644)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through exit (12-month follow-up period) for each participant. Data on adverse events were systematically collected with a "negative side effects" survey at each assessment, and at each intervention session. In addition, study personnel inquired about potential adverse events at each participant contact. All adverse events were recorded, reported, and categorized according to the funding agency, IRB, and other regulatory guidance.
Description: Definitions from study protocol:
  10.1.1 AE: Any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related.
  10.1.2 SAE Any of the following: Fatal; life-threatening; persistent/significantly disabling/incapacitating; inpatient hospitalization/prolongation of hospitalization; significant medical incident that may jeopardize the participant and requires medical/surgical intervention to prevent one of the above outcomes
Arm/Group | Mindfulness Based Therapy | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 1/385 | 3/385
Serious Adverse Events (participants affected / at risk) | 0/385 | 0/385
Other Adverse Events (participants affected / at risk) | 0/385 | 24/385
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Therapy (N=385) | Cognitive Behavioral Therapy (N=385)
Increased pain reported as associated with progressive muscle relaxation exercise (Musculoskeletal and connective tissue disorders) | 0 (0) | 24 (38) — Self-limited, mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT03115359/Prot_SAP_000.pdf